CLINICAL TRIAL: NCT06285929
Title: Community Engagement in the Development of Oncology Navigation Training
Brief Title: ACS Community Access to Resources Education and Support
Acronym: ACS CARES
Status: Enrolling by invitation | Type: Observational
Sponsor: American Cancer Society, Inc. (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Bonny Morris, Senior Director, ACS CARES, American Cancer Society, Inc.
Other Study IDs: 2013209-1
Record Dates: First submitted 2024-02-06; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Neoplasms
Keywords: Patient Navigation; Patient Satisfaction; Patient Engagement; Patient Empowerment; Patient Participation; Treatment Adherance
MeSH Terms: conditions — Neoplasms; Patient Satisfaction; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Navigated patients: Student volunteer navigation support accessing barriers to care for patients, families and caregivers with a cancer diagnosis through a social determinants of health assessment and connecting with resources with an effort to eliminate barriers.
  Interventions: Other: ACS CARES Student Navigation
- non-navigated patients: Patients, families and caregivers with a cancer diagnosis without the support of student volunteer navigation and serving as the baseline and control.
- Student volunteers: Undergraduate or graduate students volunteering with ACS CARES program to provide navigation support to patients, families and caregivers with a cancer diagnosis.
  Interventions: Other: ACS CARES Student Navigation

INTERVENTIONS:
Other: ACS CARES Student Navigation — Student volunteers providing navigation support to patients, families and caregivers with a cancer diagnosis through an SDOH assessment.
  Groups: Navigated patients; Student volunteers

SUMMARY:
The goal of this study is to evaluate the pilot phase of ACS Cares to identify key implementation outcomes and assess effectiveness of the program to improve distress, enhance communication, and reduce missed appointments and healthcare utilization.

DETAILED DESCRIPTION:
In 2023, the American Cancer Society (ACS) created a new program, ACS Cares, based on the Take the Fight experience and existing literature on non-clinical navigation. The goal of ACS Cares is to supplement existing navigation infrastructure to extend navigation services to a broader population of patients. This is accomplished through designating lower level, timely tasks to volunteers and allowing paid navigators to practice at the highest level of their license (e.g nurses proving symptom management, higher level coordination). The goal of this study is to evaluate the pilot phase of ACS Cares to identify key implementation outcomes and assess effectiveness of the program to improve distress, enhance communication, and reduce missed appointments and healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

* patients of health system's healthcare physician champions with a confirmed cancer diagnosis
* patients with a confirmed cancer diagnosis
* families of patients with a confirmed cancer diagnosis
* Caregivers of patients with a confirmed cancer diagnosis

Exclusion Criteria:

* patients, families and/or caregivers without a confirmed cancer diagnosis
* patients not receiving care from healthcare physician champions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients, families and/or caregivers with a confirmed cancer diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure the impact of ACS CARES on patient-reported outcomes: SDOH barriers | Baseline and 6 months into pilot
  SDOH barriers
Measure the impact of ACS CARES on patient-reported outcomes: Information Needs | Baseline and 6 months into pilot
  Information Needs
Measure the impact of ACS CARES on patient-reported outcomes: Distress needs | Baseline and 6 months into pilot
  Distress needs
Measure the impact of ACS CARES on patient-reported outcomes: Satisfaction with program | Baseline and 6 months into pilot
  Satisfaction with program
Measure the impact of ACS CARES on patient-reported outcomes: Unmet needs | Baseline and 6 months into pilot
  Unmet needs
Measure the impact of ACS CARES on patient-reported outcomes: Patient-provider communication | Baseline and 6 months into pilot
  Patient-provider communication
Measure the impact of ACS CARES on patient-reported outcomes: clinical trials knowledge | Baseline and 6 months into pilot
  clinical trials knowledge
Measure the impact of ACS CARES on patient-reported outcomes: Patient activation | Baseline and 6 months into pilot
  Patient activation
Measure the impact of ACS CARES on patient-reported outcomes: Financial toxicity | Baseline and 6 months into pilot
  Financial toxicity
Measure the impact of ACS CARES on patient-reported outcomes: Quality of life | Baseline and 6 months into pilot
  Quality of life
Context, Training, and Process Measures: Service Penetrance and Process Measures: Service Penetrance | through study completion, an average of 1 year
  • # of patients/caregivers approached for ACS CARES Median and range per volunteer • # of patients/caregivers who decline by refusal reason • # of patients/caregivers supported by ACS CARES Median and range per volunteer • # of patients/caregivers who received psychosocial distress screening Median and range per ACS CARES volunteer • # of patients/caregivers who received an SDOH screening Median and range per ACS CARES volunteer • # of follow-ups conducted Median and range per ACS CARES volunteer • # of in-person visits conducted Median and range per ACS CARES volunteer • # of shifts completed Median and range per ACS CARES volunteer • # of referrals received from health system team members

SECONDARY OUTCOMES:
Sociodemographic differences between ACS CARES supported and non-ACS CAREs supported patients | baseline and 1 year
  Patient characteristics: age, sex, gender (if available), race, ethnicity, insurance status, zip code, urban or rural residence, Area Deprivation Index category, and distance from cancer center (<30 minutes, 30-60 minutes, >60 minutes)
Impact of ACS CARES on treatment adherence and healthcare | baseline and 1 year
  Cancer and treatment characteristics: cancer type, date of diagnosis, type of current treatment (Surgery, Chemotherapy, Radiation Therapy, Targeted Therapy, Immunotherapy, Stem Cell or Bone Marrow Transplant, Hormone Therapy), total clinic appointments, # clinic appts missed/cancelled, total infusion appointments, # infusion appointments missed/cancelled, total radiation treatment appts, # radiation treatment appointments missed/cancelled, enrolled in a clinical trial (y/n), start date of clinical trial participation, ER visits, hospitalizations, ICU admissions, total cost of care. For new patients during baseline or intervention time periods, date of first clinic visit.
Context, Training, and Process Measures: Volunteer Satisfaction | 1 year
  Volunteer Satisfaction Index

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA Health, Los Angeles, California
  - American Cancer Society, Kennesaw, Georgia
  - University of Iowa Health Care, Iowa City, Iowa
  - Medical University Hospital Authority, Hollings Cancer Center, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided